CLINICAL TRIAL: NCT01243827
Title: Comparison of Effect of cARvedilol Compared To bISoprolol on cenTral Pulse Pressure in Hypertension (ARTIST) Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yoshio Matsui (Other)
Responsible Party: Sponsor-Investigator, Yoshio Matsui, Sponsor investigator, Jichi Medical University
Organization: Jichi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTIST
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2010-11

CONDITIONS: Hypertension
Keywords: Hypertension, carvedilol, bisoprolol, central pulse pressure, pulse pressure amplification, reflection magnitude, LV mass index, LV diastolic function
MeSH Terms: conditions — Hypertension | interventions — Carvedilol; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carvedilol (Experimental): carvedilol is administered after randomization at a dose of 10 mg once daily, and if needed, titrated to 15 mg and to a maximum of 20 mg to achieve a clinic BP <140/90 mmHg.
  Interventions: Drug: carvedilol
- bisoprolol (Experimental): bisoprolol is administered after randomization at a dose of 2.5 mg once daily, and if needed, titrated to 3.75 mg and to a maximum of 5.0 mg to achieve a clinic BP <140/90 mmHg.
  Interventions: Drug: bisoprolol

INTERVENTIONS:
Drug: carvedilol — carvedilol is administered after randomization at a dose of 10 mg once daily, and if needed, titrated to 15 mg and to a maximum of 20 mg to achieve a clinic BP <140/90 mmHg.
  Arms: carvedilol
Drug: bisoprolol — bisoprolol is administered after randomization at a dose of 2.5 mg once daily, and if needed, titrated to 3.75 mg and to a maximum of 5.0 mg to achieve a clinic BP <140/90 mmHg.
  Arms: bisoprolol

SUMMARY:
The purpose of this study is to compare of carvedilol, a vasodilating beta-blocker and bisoprolol, a beta1- selective beta-blocker for reducing the central pulse pressure and thereby left ventricular (LV) mass in never-treated hypertensive patients.

DETAILED DESCRIPTION:
Carvedilol and bisoprolol are established beta-blockers for treating hypertension or chronic heart failure because these beta-blockers have cardio-protective effects. Recent studies have shown that the change in central pulse pressure is more closely associated with the change in cardiac load than the change in brachial pressure during hypertension treatment. Vasodilating beta-blockers may decrease central pulse pressure more than beta1- selective beta-blockers, because vasodilators reduced the magnitude of reflection wave by dilating peripheral muscular arteries. The investigators hypothesized that carvedilol, a vasodilating beta-blocker, would be more effective than bisoprolol, a beta1- selective beta-blocker in reducing central pulse pressure and thereby LV mass, through the reduction in the magnitude of reflection wave. The aim of the present study was to test this hypothesis in an active controlled, 2-arm parallel group comparison, prospective randomized open blinded end-point (PROBE) design study. At least 100 patients will be enrolled in each group and the follow up duration will be 48 weeks. The primary endpoint is to compare the change in central pulse pressure between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Never-treated hypertensive subjects, aged 20-80 years (at the time of informed consent), regardless of sex
* Clinic systolic BP/diastolic BP > 140/90 mmHg in a sitting position.

Exclusion Criteria:

* Beta-blocker contraindications(asthma, COPD…)
* Heart rate less than 55 bpm
* Subjects treated with nitrates
* Grade 3 hypertension (≥180 and/or ≥110 mmHg)
* Secondary hypertension or malignant hypertension
* History of heart failure, coronary artery disease, and stroke
* Arrhythmia
* Renal dysfunction (serum creatinine ≥2.0 mg/dl)
* Hepatic dysfunction (AST and/or ALT ≥100 IU/l)
* A history of or a suspected malignant tumor within 5 years of enrollment
* Chronic inflammatory disease
* Pregnancy, childbearing potential with inadequate contraception, breast feeding
* Inability to give informed consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change in central pulse pressure (pulse pressure amplification) | 12 months

SECONDARY OUTCOMES:
Change in LV mass index Changes in LV diastolic functions (E/Em, left atrium volume) Changes in urinary albumin excretion, B-type natriuretic peptide (BNP), HOMA-IR, and oxidative stress (urinary 8-isoprostane). Change in ambulatory BP | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuomi Kario, Principal Investigator — Jichi Medical University
Locations (1):
- Iwakuni City Medical Center, Yamaguchi, Japan